CLINICAL TRIAL: NCT02317068
Title: Increasing Atrial Base Rate Pacing to Reduce Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chancellor of research, Vice-Chancellor for Research in UMSU, Urmia University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMSU-Cardiology-4
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Sick Sinus Syndrome; Paroxysmal Atrial Fibrillation
Keywords: sick sinus syndrome; paroxysmal atrial fibrillation; atrial pacing; high atrial base rate pacing
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Atrial Base Rate Pacing (Experimental): The base rate of pacemaker will be determined 75-100 beats/minute in condition that during first step of follow-up, his/her atrial pacing will be more than 80% of atrial high rate/automatic mode switch
  Interventions: Device: HBR
- Device Default (Active Comparator): The base rate of pacemaker will be determined 60 beats/minute
  Interventions: Device: DD

INTERVENTIONS:
Device: HBR
  Other Names: High Atrial Base Rate Pacing
  Arms: High Atrial Base Rate Pacing
Device: DD
  Other Names: Device Default
  Arms: Device Default

SUMMARY:
This study aims to determine whether increasing atrial base rate pacing to achieve at least 75-80% atrial pacing in patients with sick sinus syndrome undergoing the implementation of dual-chamber pacemaker can be useful to prevent or decrease the atrial fibrillation during 6 months follow-up duration.

ELIGIBILITY:
Inclusion Criteria:

* Sick sinus syndrome patients having dual-chamber pacemaker
* Having paroxysmal AF defined as at least 2 episodes of AHR/AMS >190 b/min lasting >6 minutes
* Having normal atrioventricular conduction

Exclusion Criteria:

* Other clinical indications for pacing except sick sinus syndrome (bradycardia-tachycardia syndrome)
* History of acute coronary syndrome
* Significant heart valve disease
* Chronic AF before randomization
* Overt heart failure
* Malignancy
* Any reasons for antiarrhythmic medication use
* Inability to follow patients every 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Atrial high rate/Automatic mode switch episodes | During 6 Months
  The number of AHR/AMS episodes recorded by pacemaker

SECONDARY OUTCOMES:
Stroke | During 6 months
  The development of stroke during follow-up
Myocardial infarction | During 6 months
  The development of MI during follow-up confirmed by ischemic chest pain, 12-ECG, or cardiac enzyme elevation
Heart failure | During 6 months
  The development or progression of heart failure during follow-up
Worsening Functional Class | During 6 months
  The worsening of functional class
Death | During 6 months
  Death

CONTACTS AND LOCATIONS:
Locations (1):
- Seyyed-al-Shohada Heart Center, UMSU, Urmia, West Azerbaijan Province, Iran